CLINICAL TRIAL: NCT05189704
Title: The Effect of Patient-controlled Analgesia (Ketorolac vs. Fentanyl) on the Development of Postoperative Nausea and Vomiting in Patients Undergoing Microvascular Decompression: a Prospective Randomized Controlled Trial
Brief Title: The Effect of PCA on PONV After Microvascular Decompression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Koo, Assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MVD-PCA
Record Dates: First submitted 2021-12-07; First posted 2022-01-12 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Anti-Inflammatory Agents, Non-Steroidal; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSAID group (Experimental): NSAID based patient-controlled analgesia will connected to intravenous line for pain control.
  Interventions: Drug: NSAID
- Opioid group (Active Comparator): Opioid based patient-controlled analgesia will connected to intravenous line for pain control.
  Interventions: Drug: Opioid

INTERVENTIONS:
Drug: NSAID — NSAID based patient-controlled analgesia will connected to intravenous line for pain control.
  Arms: NSAID group
Drug: Opioid — Opioid based patient-controlled analgesia will connected to intravenous line for pain control.
  Arms: Opioid group

SUMMARY:
This study is a randomized, controlled, double-blinded, and parallel design study. A total 94 patients will be randomized to receive ketorolac or fentanyl based patient-controlled analgesia after microvascular decompression surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo elective microvascular decompression surgery
* American Society of Anesthesiologists grade 1 or 2
* 19 - 65 years old

Exclusion Criteria:

* Refuse to participate to the study
* Refuse to use Patient-controlled analgesia
* Body Mass Index < 18.5 kg/m2 or > 35 kg/m2
* history of craniotomy or chemotheraphy
* Patients who used preoperative antiemetics within 24h before surgery
* Severe renal or hepatic dysfunction
* Pregnant

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | postoperative 48 hours
  Incidence

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | Postoperative 30 minutes, 1 hours, 24 hours, 48 hours
  Severity accessed using numeric rating scale (0=none, 10=worst PONV possible)
Postoperative pain | Postoperative 30 minutes, 1 hours, 24 hours, 48 hours
  pain intensity will be assessed using numeric rating scale (0=none, 10=worst pain possible)
Postoperative PCA consumption | Postoperative 30 minutes, 1 hours, 24 hours, 48 hours
Rescue antiemetics requirement | Postoperative 30 minutes, 1 hours, 24 hours, 48 hours
Rescue analgesic requirement | Postoperative 30 minutes, 1 hours, 24 hours, 48 hours
Satisfaction score for postoperative nausea and vomiting | postoperative 48 hours
  using 11-point scale (0=Worst dissatisfied, 10=Very satisfied)
Satisfaction score for postoperative pain | postoperative 48 hours
  using 11-point scale (0=Worst dissatisfied, 10=Very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Koo, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No